CLINICAL TRIAL: NCT01530074
Title: Quantitative Sensory Testing of the Lower Lip After Inferior Alveolar Nerve Block, and Evaluation of the Role of the Contra-lateral Inferior Alveolar Nerve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: we have not succeeded in recruiting patients
Sponsor: K Blal (Other)
Responsible Party: Sponsor-Investigator, K Blal, Dr. Blal Kifah, Hadassah Medical Organization
Organization: Hadassah Medical Organization (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: QSensory-HMO-CTIL
Record Dates: First submitted 2012-02-07; First posted 2012-02-09 (Estimated); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Healthy
Keywords: Mandibular nerve; Mental nerve; Mandibular incisive nerve; Local anesthesia; None, only healthy subjects will be enrolled in this study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Procedure: Temporary blocking of mandibular nerve

INTERVENTIONS:
Procedure: Temporary blocking of mandibular nerve — IM. Lidocaine 2% 7.2ML

SUMMARY:
The purpose of this study is to determine the contribution of the innervation of the contra-lateral mandibular nerve for the innervation of the lower lip area.

The investigators hypothesis is that the sensation of the lower lip is contributed by both mandibular nerves (from both sides of the jaw).

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no systemic diseases, chronic medication, past nerve injury, or sensory complaint.

Exclusion Criteria:

* Hypersensitivity/allergy to local anesthetic materials
* Systemic diseases, Chronic medication
* Past nerve injury
* Congenital or acquired deformity in the lower jaw
* Past fractures/neoplasm of the lower jaw
* Past surgery to the lower lip

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-08 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Quantitative sensory test | 15 minutes
  Measurement of sensory conduction of A-beta, A-delta, C-fibers of mandibular nerve, using electronic neurometer.